CLINICAL TRIAL: NCT06021236
Title: Efficacy of a Mindfulness-Based Intervention on Resilience, Perceived Stress, Anxiety, and Depression, in Patients With Cardiovascular Implantable Electronic Device: A Mixed-Methods Research
Brief Title: Efficacy of a Mindfulness-Based Intervention in Patients With Cardiovascular Implantable Electronic Device
Acronym: MBI-CIED
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Chien Chih-Yin (Other)
Collaborators: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Sponsor-Investigator, Chien Chih-Yin, Director, National Taipei University of Nursing and Health Sciences
Organization: National Taipei University of Nursing and Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MKC-23MMHIS220e; 23MMHIS220e (Registry Identifier: CYChien)
Record Dates: First submitted 2023-06-29; First posted 2023-09-01 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Mindfulness Training; Cardiac Resynchronization Therapy Devices; Resilience, Psychological; Anxiety; Depression; Perceived Stress
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: This study is a randomized clinical trial design (randomized clinical trial) with qualitative analysis, which is a mixed-methods research. Research objects were randomly assigned to the experimental and control groups in a 1:1 manner. The experimental group received the mindfulness-based intervention designed and routine care, and the control group received usual care. A total of four questionnaires were filled in the pretest (T0), the first month of discharge (T1), the 3rd month of discharge(T2), and the 6th month of discharge (T3), including anxiety, depression, mental toughness, and stress perception. Qualitative interviews were conducted at T2 and T3 to understand the improvement of psychological problems.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mindfulness-based intervention and routine care (Experimental): mindfulness-based intervention including: breathing awareness, body scanning, mindful yoga, mindful eating, and loving-kindness meditation. From the time when the patients signed up to be the first to receive the cardiac device surgery schedule, the experimental group that met the including criteria, in addition to following the routine care of the hospital, was involved in teaching the above mindfulness skills, and Osaka continued to follow the regular care.
  Interventions: Behavioral: mindfulness-based intervention; Other: CIED procedure routine care
- The control group received the CIED procedure routine care (Other): From the time when the patients signed up to be the first to receive the cardiac device surgery schedule, the control group that met the including criteria take routine care of the hospital.
  Interventions: Other: CIED procedure routine care

INTERVENTIONS:
Behavioral: mindfulness-based intervention — Diet meditation breath awareness body scan mindfulness yoga Compassionate blessing
  Other Names: mindfulness-based intervention with CIED procedure routine care
  Arms: mindfulness-based intervention and routine care
Other: CIED procedure routine care — CIED procedure home care guidance

SUMMARY:
An implantable cardiac defibrillator (implantable cardioverter-defibrillator; ICD) can effectively improve heart rhythm problems and reduce sudden death, and is widely used in the treatment of high-risk patients with fatal arrhythmias or heart rhythm problems that cannot be controlled by drugs . In the whole case of arrhythmia, after receiving home-based cardiac fibrillator treatment, Patients often experience uncertainty, feel the changes in heart, feel the shock of being shocked by the electric shock, and worry about death, These psychological distress, which were characterized by anxiety and depression. for universal. About 25% of patients present with symptoms of anxiety at the time of hospitalization, and 50% suffer from depression which seriously affects quality of life. Therefore, the main purpose of this study to alleviate the occurrence of anxiety and depression, promote disease patients to regain life adaptation, develop accessible care strategies with midfulness-based intervention to help patients overcome psychological distress, reduce stress, anxiety and prevent depression.

DETAILED DESCRIPTION:
This study with randomized clinical trial design (randomized clinical trial) and qualitative research, which is a qualitative mixed-methods research. Patients were randomly assigned to the experimental group and the control group in a 1:1 manner. The experimental group received the mindfulness-based intervention designed and routine care , and the control group received general routine care. Both groups completed a total of four questionnaires at the pretest (T0), discharge (T1), the first month of discharge (T2), and the third month of discharge (T3), including anxiety, depression, resilience, stress perception scale and other basic data such as demographics and disease characteristics were collected in the pretest.

This study held an expert meeting to extract the techniques of mindfulness measures suitable for this disease attribute and the elderly group, including: breathing awareness, body scanning, mindful yoga, mindful eating, and loving-kindness meditation. From the time when the patient signed up for the first cardiac device surgery schedule, the experimental group who met the including criteria followed the routine care of the hospital and was involved in teaching the above mindfulness skills, while the control group still followed the routine care.

ELIGIBILITY:
Inclusion Criteria:

1. Patients receiving implanted cardiac devices for the first time (including cardiac defibrillator ICD and Pacemaker).
2. Adults over 20 years old.
3. Those who have clear consciousness and can communicate in Chinese and Taiwanese.
4. Score of 8 or above on the Hospital Anxiety or Depression Scale.
5. Barthel Index above 70 points.

Exclusion Criteria:

1. Diagnosed with dementia by a physician.
2. Diagnosed with mental disorders, including cognitive disorders, organic psychosis and affective psychosis.
3. Patients who have been diagnosed with cancer.
4. Long-term bed ridden.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety | From enrollment to the end of treatment at 6 months
  This study used the Hospital Anxiety and Depression Scale (HADS) to assess anxiety in patients. This scale provides anxiety (HADS-A) scores.
Resilience | From enrollment to the end of treatment at 6 months
  This study uses the Connor-Davidson Resilience Scale (Connor-Davidson Resilience Scale), which was developed by Connor and Davidson (2003) in the United States who regarded resilience as a measurable stress response ability.
Perceived Stress | From enrollment to the end of treatment at 6 months
  This study uses the Perceived Stress Scale, which was compiled by Cohen et al. (1983) and translated from the Chinese version of Chu and Gao (2005). , the degree of stress in life.
Depression | From enrollment to the end of treatment at 6 months
  This study used the Hospital Anxiety and Depression Scale (HADS) to assess depression in patients. This scale provides anxiety (HADS-D) scores.

SECONDARY OUTCOMES:
Demographic Information | From enrollment to the end of treatment at 6 months
  Collect age, gender, education level, marital status, occupation, smoking, drinking, disease history, other disease history, and exercise habits with self-made basic data sheets.
body mass index | From enrollment to the end of treatment at 6 months
  weight and height will be combined to report BMI in kg/m^2
Feelings and experiences by interview of home-based cardiac device patients receiving pre-procedure mindfulness intervention program | From enrollment to the end of treatment at 6 months
  Intentional sampling with phenomenological method. Conduct one-on-one interview recordings for the research subjects in the experimental group to collect the feelings and experiences of patients with implanted cardiac devices who received the mindfulness-based preoperative intervention program. It is expected to close the case until the data is saturated.

CONTACTS AND LOCATIONS:
Overall Officials: CY Chien, PI, Study Chair — MKC/MMH
Locations (1):
- MacKay Junior College of Medicine, Nursing and Management, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
The research data belongs to the researcher and is expected to be destroyed after 2 years

REFERENCES:
- [Result] Freedenberg VA, Thomas SA, Friedmann E. A pilot study of a mindfulness based stress reduction program in adolescents with implantable cardioverter defibrillators or pacemakers. Pediatr Cardiol. 2015 Apr;36(4):786-95. doi: 10.1007/s00246-014-1081-5. Epub 2014 Dec 12. PMID 25519914
- [Result] Hazlett-Stevens H, Singer J, Chong A. Mindfulness-Based Stress Reduction and Mindfulness-Based Cognitive Therapy with Older Adults: A Qualitative Review of Randomized Controlled Outcome Research. Clin Gerontol. 2019 Jul-Sep;42(4):347-358. doi: 10.1080/07317115.2018.1518282. Epub 2018 Sep 11. PMID 30204557
- [Result] Hopgood DA, Czosek RJ, Bakas T, Garritano N, Gillespie GL. The Capture Gap: Implantable Cardioverter-Defibrillator Quality of Life. Clin Nurs Res. 2020 Feb;29(2):97-107. doi: 10.1177/1054773818803741. Epub 2018 Oct 7. PMID 30295057
- [Result] Li SYH, Bressington D. The effects of mindfulness-based stress reduction on depression, anxiety, and stress in older adults: A systematic review and meta-analysis. Int J Ment Health Nurs. 2019 Jun;28(3):635-656. doi: 10.1111/inm.12568. Epub 2019 Jan 17. PMID 30656813
- [Result] Marino F, Failla C, Carrozza C, Ciminata M, Chila P, Minutoli R, Genovese S, Puglisi A, Arnao AA, Tartarisco G, Corpina F, Gangemi S, Ruta L, Cerasa A, Vagni D, Pioggia G. Mindfulness-Based Interventions for Physical and Psychological Wellbeing in Cardiovascular Diseases: A Systematic Review and Meta-Analysis. Brain Sci. 2021 May 29;11(6):727. doi: 10.3390/brainsci11060727. PMID 34072605
- [Result] Rafsanjani MHAP, Masoudi S, Radmanesh M, Bostani Z. Comparison of depression and anxiety among pacemaker and implantable cardioverter-defibrillator recipients: A cross-sectional study. Pacing Clin Electrophysiol. 2021 Feb;44(2):235-239. doi: 10.1111/pace.14152. Epub 2021 Jan 12. PMID 33372277
- [Result] Schulz SM, Ritter O, Zniva R, Nordbeck P, Wacker C, Jack M, Groschup G, Deneke T, Puppe F, Ertl G, Angermann C, Stork S, Pauli P. Efficacy of a web-based intervention for improving psychosocial well-being in patients with implantable cardioverter-defibrillators: the randomized controlled ICD-FORUM trial. Eur Heart J. 2020 Mar 14;41(11):1203-1211. doi: 10.1093/eurheartj/ehz134. PMID 30957867